CLINICAL TRIAL: NCT00001579
Title: A Phase I Trial of 5-Fluorouracil Given With 776C85 (GW776) and Low-Dose Leucovorin in Adult Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 970136; 97-C-0136
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2006-07-17 (Estimated); Status verified 2000-05

CONDITIONS: Lymphoma; Neoplasms
Keywords: Biochemical Modulation; Dihydropyrimidine Dehydrogenase; Oral Administration; Pharmacokinetics
MeSH Terms: conditions — Lymphoma; Neoplasms | interventions — Fluorouracil; eniluracil; Leucovorin

INTERVENTIONS:
Drug: 5-Fluorouracil
Drug: Ethynyluracil
Drug: Leucovorin

SUMMARY:
This is a dose escalation study.

During the first period of this study, an initial pharmacological assessment of fluorouracil administered intravenously along with oral leucovorin calcium is made. Leucovorin calcium is given orally bid on days 1-3. Fluorouracil is given as a 24 hour infusion on day 2.

After a 2 week rest period and resolution of any toxicities experienced during the first period of treatment, patients are given an escalating dose of fluorouracil with fixed doses of leucovorin calcium and ethynyluracil. Ethynyluracil and leucovorin calcium are given bid orally on days 1-3 of each week. Fluorouracil is given bid orally on day 2 of each week. Treatment is repeated for three weeks followed by a one week rest period.

3 to 6 patients are enrolled at each dose level. Dose escalation proceeds until the maximum tolerated dose (MTD) is determined. MTD is defined as the dose preceding that at which 2 or more patients experience dose limiting toxicity.

DETAILED DESCRIPTION:
The primary purpose of this Phase I protocol is to develop an orally administered regimen of fluorouracil (5-FU) given with fixed doses of leucovorin (LV) and 776C85 (GW776), a mechanism-based inhibitor of dihydropyrimidine dehydrogenase (DPD), the rate-limiting enzyme involved in the catabolism of 5-FU. In the presence of 776C85, 5-FU is cleared by renal mechanisms. The schedule employed is intended to mimic the pharmacologic profile associated with a 24 hour weekly continuous infusion of 5-FU without the need for an indwelling central venous catheter. The target population is adult cancer patients with solid tumors.

The first week, each patient will receive a single dose of 5-FU given by 24 hour continuous IV infusion at its recommended Phase II dose with low-dose oral LV. In the third week, the patient will begin 776C85 (GW776) and LV PO on days 1, 2, 3 at fixed doses. Oral 5-FU will be given on day 2, and the dose will be escalated in successive cohorts of patients. Treatment will be repeated weekly for three weeks, followed by a one week break. The dose of 5-FU will be adjusted according to individual tolerance. Cohorts of three patients will be entered at each dose level of 5-FU, which will be escalated until dose-limiting toxicity is seen (guidelines are outlined in the following schema). Treatment will be continued indefinitely until evidence of disease progression, provided the patient is tolerating therapy and wishes to continue.

Biochemical monitoring suggests that there is profound and sustained inhibition of DPD with a single dose of 20 mg PO 776C85 days 1-3 each week for three of four weeks. Once the MTD has been defined for the once daily dosing on days 1, 2, 3 schedule, a simplified schedule will be evaluated in which a single dose of 776C85 on day 1 in the evening, with oral leucovorin days 1 and 2, and 5-FU given day 2 as a single dose.

Since the pharmaceutical company has decided to go with a combined tablet of eniluracil/5-FU for future studies, the new schedule will be oral leucovorin on days 1 & 2, with 776C85 and 5-FU both given day 2 as a single dose.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Histologically proven solid tumor that has failed standard therapy or for which no such therapy exists.

Tumor may be locally advanced and unresectable, recurrent and/or metastatic.

Lymphomas with minimal or no involvement of bone marrow are also eligible.

No primary malignancies or metastatic disease of the CNS.

No symptomatic pre-existing peripheral neuropathy.

PRIOR/CURRENT THERAPY:

BIOLOGIC THERAPY:

No immunotherapy within past 4 weeks.

Recovered from toxic effects.

CHEMOTHERAPY:

No chemotherapy within past 4 weeks (6 weeks for nitrosoureas).

No mitomycin within past 12 weeks.

Recovered from toxic effects.

ENDOCRINE THERAPY: Not specified.

RADIOTHERAPY:

No radiotherapy within past 2 weeks (8 weeks for strontium therapy).

Recovered from toxic effects.

SURGERY: Recovered from prior surgery.

OTHER: No concurrent cimetidine.

PATIENT CHARACTERISTICS:

AGE: 18 and over.

PERFORMANCE STATUS: ECOG 0-2.

LIFE EXPECTANCY: Not specified.

HEMATOPOIETIC:

Absolute granulocyte count at least 2000/mm(3);

Platelet count at least 100,000/mm(3).

HEPATIC:

Bilirubin no greater than 2 times upper normal limit;

SGOT/SGPT no greater than 4 times upper normal limit.

RENAL:

Creatinine no greater than 1.6 mg/dL;

Creatinine clearance greater than 55 mL/min.

OTHER:

Not pregnant or nursing.

Fertile patients must use effective contraception.

Not HIV positive.

No active infections requiring intravenous antibiotic therapy.

No other serious concurrent illness.

No evidence of hemolytic uremic syndrome.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 1997-06; Study Completion 2001-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Evans RM, Laskin JD, Hakala MT. Assessment of growth-limiting events caused by 5-fluorouracil in mouse cells and in human cells. Cancer Res. 1980 Nov;40(11):4113-22. No abstract available. PMID 6162543
- [Background] Spears CP, Shani J, Shahinian AH, Wolf W, Heidelberger C, Danenberg PV. Assay and time course of 5-fluorouracil incorporation into RNA of L1210/0 ascites cells in vivo. Mol Pharmacol. 1985 Feb;27(2):302-7. PMID 2578605
- [Background] Calabro-Jones PM, Byfield JE, Ward JF, Sharp TR. Time-dose relationships for 5-fluorouracil cytotoxicity against human epithelial cancer cells in vitro. Cancer Res. 1982 Nov;42(11):4413-20. No abstract available. PMID 7127282